CLINICAL TRIAL: NCT06601478
Title: Development and Implementation of a Tool for the Evaluation and Monitorization of Mediterranean Lifestyle At Clinical Settings: MEDLIFE Index, a Proof of Concept Study
Brief Title: Development and Implementation of a Tool for the Evaluation and Monitoring of the Mediterranean Lifestyle in the Clinical Setting
Acronym: MedLIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Hospital Universitario Juan Ramón Jiménez (Unknown)
Responsible Party: Principal Investigator, Mercedes Sotos Prieto, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNS2022-135623
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-09

CONDITIONS: Lifestyle
Keywords: Lifestyle behaviours; Cardiovascular disease; Cardiovascular event; Intervention; Health App; Prevention; Mediterranean Diet
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The intervention group will complete de MEDLIFE questionnaire and use the MEDLIFE online app where they will receive counselling on lifestyle, food choices or physical activity. Meanwhile, the control group will only complete the MEDLIFE questionnaire, but will not receive the app lifestyle intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle Intervention (Experimental): Participants will undergo the MEDLIFE evaluation and will talk over their results and recommendations with the health care providers (cardiologists, nurses or dietitians) to improve habits identified as inadequate.
  The intervention group will obtain access to the MEDLIFE online app and will receive personal text messages based on the MEDLIFE test to improve each of the items included in the tool. The available resources will be based on the recommendations for diet, physical activity, sleep and social interaction.
  At the beginning and in each of the 4 visits, the following determinations will be done in both groups: anthropometric and biochemical measurements by trained stuff, arterial pressure, MEDLIFE scoring, sociodemographic questions, several questionnaires, and other relevant information obtained from medical histories.
  Interventions: Behavioral: The MedLIFE app
- Control, no Lifestyle Intervention (No Intervention): Participants will undergo the MEDLIFE evaluation and will talk over their results and recommendations with the health care providers (cardiologists, nurses or dietitians) to improve habits identified as inadequate.
  The control group will continue with their current lifestyle and will receive a handout with lifestyle recommendations.
  At the beginning and in each of the 4 visits, the following determinations will be done in both groups: anthropometric and biochemical measurements by trained stuff, arterial pressure, MEDLIFE scoring, sociodemographic questions, several questionnaires, and other relevant information obtained from medical histories.

INTERVENTIONS:
Behavioral: The MedLIFE app — The intervention arm will receive the lifestyle counselling by the MEDLIFE app, and the control arm will go on with standard lifestyle recommendations in the form of a two-page written handout.
  Arms: Lifestyle Intervention

SUMMARY:
The main goal is to develop a health online app based on a Mediterranean lifestyle score (diet, cooking preferences, rest, physical activity, social habits, conviviality) and its implementation in clinical settings with patients that have suffered from a cardiovascular event. This is a pilot study that will allow an integral assessment of health as an attempt to decrease obesity, one of the main risk factors of cardiovascular disease, as well as to improve the prevention of secondary events.

The main goal involves the following specific objectives:

Developing and transferring the previously validated questionnaire in Spanish population (MEDLIFE index, MEDiterranean LIFEstyle) to evaluate adherence to a Mediterranean lifestyle an online app, that allows:

To evaluate and to monitor the adherence to the MEDLIFE throughout time.

To use the MEDLIFE online app to obtain customized recommendations according to the results (an instantaneous generation of a resume of results).

To start conversations between patient and health workers to improve patient's lifestyles, obesity or related parameters and cardiovascular health.

To keep information in a safe way that will allow it to be linked to other health indicators.

Conducting a qualitative study using personal interviews with health providers and patients, to evaluate acceptation, feasibility, barriers, or limitations when using the MEDLIFE app in clinical practice, aiming for the app's enhancing.

Conducting a pilot study of implementation of MEDLIFE in clinical settings, in patients with a cardiovascular event (myocardial infarction, ictus, angina, ischemic cardiopathy) (n= 80-100, trying parity between men and women).

This is the project's intervention part.

To evaluate changes in MEDLIFE and its components, anthropometric and biochemical measurements between baseline, 3-month, 6-month and 8-month follow-up.

Following participants by means of revision of medical reports and clinical histories to register future cardiovascular events (dynamic).

DETAILED DESCRIPTION:
Participants will be selected from the clinical cardiology and cardiac rehabilitation or internal medicine services. Each physician will recruit patients from among those assigned to his or her practice, just as they are discharged from the hospital after a cardiovascular event.

The online application will be suitable for tablet, mobile and web use. For its development, a specialist web/app development company will be contracted and will follow the indications of the research team.

The application, visually attractive, should allow a quick and easy evaluation of MEDLIFE and, in addition, include interactive features that raise awareness and motivate users to change their health habits. Thus, when the participant has completed the questionnaire, a results page will be automatically generated with a color scale to indicate what needs to be improved (red, indicating a factor to be considered for improvement; green, the recommendations are met and the participant is performing adequately). Also, specific recommendations will be provided to achieve the objectives of those factors that can be improved. In this way, the results will be ready to be evaluated and discussed with the healthcare professional. The design of the app will be inclusive to allow the use of the app by people with certain disabilities (it will allow the questions to be read by a voice (audio), for people with disabilities, vision loss or illiterate). This objective will be carried out with the help of a computer technician specialized in the development of mobile applications and web pages.

In addition, physicians will be able to monitor their patients at each visit, entering themselves the data obtained from MEDLIFE as well as anthropometric and analytical parameters. All this information entered into the app will be available for research use by the researchers for the project, in an anonymized form.

The data will be stored in a secure, password-protected Firebase system to allow data analysis and tracking. A consent, medical disclaimer and privacy policy will be included in the app.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years and below 75 years.
* Absence of language barriers
* To be included in the cardiac rehabilitation programme
* Capacity to comprehend, and answer the questionnaires, as well as to sign the informed consent.
* Being a Spanish resident for a period of at least 1 year prior to the beginning of the study.
* Not planning to permanently reside outside of Spain within the year.
* Having suffered from a cardiovascular event (myocardial infarction, ictus, angina, ischemic cardiopathy).

Exclusion Criteria:

* Limitation to adhering to the recommendations.
* Severe risk factors and/or with complicated control.
* Chronic diseases not related to coronary disease (severe mental illness, congenital, susceptible to decompensation endocrinopathies, and gastrointestinal diseases with diarrhoea).
* Patients that have an alternative private health insurance that doesn´t allow an electronic access to their data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Mediterranean Lifestyle Index (MedLIFE) | 6-8 months
  The primary outcome will be an increased adherence to the MedLIFE Index (0-28 points), indicating better adherence to the Mediterranean lifestyle. Participants in the intervention group will aim to enhance diet quality with moderate caloric restriction, engage in at least 150 minutes of moderate-intensity physical activity weekly, sleep 6-8 hours nightly with naps as needed, and increase resilience through positive social connections to manage stress.
Changes in intermediate lipid biomarkers of CVD | 6-8 months
  Changes in cardiovascular disease biomarkers measured through blood and urine tests:
  * Total cholesterol mg/dL
  * Low-density lipoprotein cholesterol mg/dL
  * Non-high-density, cholesterol mg/dL
  * High -density lipoprotein cholesterol mg/dL
  * Apolipoprotein B mg/dL
  * Triglycerides mg/dL
  * Remnant cholesterol mg/dL
  * Lipoprotein(a) mg/dL
  * Fraction of lipoprotein(a) mg/dL
Changes in intermediate biomarkers of CVD: blood pressure | 6-8 months
  Changes in blood pressure, other biomarkers of CVD:
  * Systolic blood pressure (mmHg)
  * Diastolic blood pressure (mmHg)
Changes in intermediate biomakers of CVD: glucose metabolism | 6-8 months
  Changes in glycated hemoglobin %
Changes in anthropometric metrics: hip and waist circunference (cm) | 6-8 months
  Changes in:
  * Hip circunference (cm)
  * Waist circunference (cm)
Changes in anthropometric metrics: BMI | 6-8 months
  Body mass index (BMI): measured by weight (Kg) and height (m²) combined

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Juan Ramón Jiménez, Huelva, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernaez A, Zomeno MD, Degano IR, Perez-Fernandez S, Goday A, Vila J, Civeira F, Moure R, Marrugat J. Excess Weight in Spain: Current Situation, Projections for 2030, and Estimated Direct Extra Cost for the Spanish Health System. Rev Esp Cardiol (Engl Ed). 2019 Nov;72(11):916-924. doi: 10.1016/j.rec.2018.10.010. Epub 2018 Nov 23. English, Spanish. PMID 30473259
- [Background] Williamson EJ, Walker AJ, Bhaskaran K, Bacon S, Bates C, Morton CE, Curtis HJ, Mehrkar A, Evans D, Inglesby P, Cockburn J, McDonald HI, MacKenna B, Tomlinson L, Douglas IJ, Rentsch CT, Mathur R, Wong AYS, Grieve R, Harrison D, Forbes H, Schultze A, Croker R, Parry J, Hester F, Harper S, Perera R, Evans SJW, Smeeth L, Goldacre B. Factors associated with COVID-19-related death using OpenSAFELY. Nature. 2020 Aug;584(7821):430-436. doi: 10.1038/s41586-020-2521-4. Epub 2020 Jul 8. PMID 32640463
- [Background] Esposito K, Kastorini CM, Panagiotakos DB, Giugliano D. Mediterranean diet and metabolic syndrome: an updated systematic review. Rev Endocr Metab Disord. 2013 Sep;14(3):255-63. doi: 10.1007/s11154-013-9253-9. PMID 23982678
- [Background] InterAct Consortium; Romaguera D, Guevara M, Norat T, Langenberg C, Forouhi NG, Sharp S, Slimani N, Schulze MB, Buijsse B, Buckland G, Molina-Montes E, Sanchez MJ, Moreno-Iribas MC, Bendinelli B, Grioni S, van der Schouw YT, Arriola L, Beulens JW, Boeing H, Clavel-Chapelon F, Cottet V, Crowe FL, de Lauzon-Guillan B, Franks PW, Gonzalez C, Hallmans G, Kaaks R, Key TJ, Khaw K, Nilsson P, Overvad K, Palla L, Palli D, Panico S, Quiros JR, Rolandsson O, Romieu I, Sacerdote C, Spijkerman AM, Teucher B, Tjonneland A, Tormo MJ, Tumino R, van der AD, Feskens EJ, Riboli E, Wareham NJ. Mediterranean diet and type 2 diabetes risk in the European Prospective Investigation into Cancer and Nutrition (EPIC) study: the InterAct project. Diabetes Care. 2011 Sep;34(9):1913-8. doi: 10.2337/dc11-0891. Epub 2011 Jul 25. PMID 21788627
- [Background] Esposito K, Maiorino MI, Bellastella G, Chiodini P, Panagiotakos D, Giugliano D. A journey into a Mediterranean diet and type 2 diabetes: a systematic review with meta-analyses. BMJ Open. 2015 Aug 10;5(8):e008222. doi: 10.1136/bmjopen-2015-008222. PMID 26260349
- [Background] Echeverria G, McGee EE, Urquiaga I, Jimenez P, D'Acuna S, Villarroel L, Velasco N, Leighton F, Rigotti A. Inverse Associations between a Locally Validated Mediterranean Diet Index, Overweight/Obesity, and Metabolic Syndrome in Chilean Adults. Nutrients. 2017 Aug 11;9(8):862. doi: 10.3390/nu9080862. PMID 28800091
- [Background] Sotos-Prieto M, Bhupathiraju SN, Mattei J, Fung TT, Li Y, Pan A, Willett WC, Rimm EB, Hu FB. Changes in Diet Quality Scores and Risk of Cardiovascular Disease Among US Men and Women. Circulation. 2015 Dec 8;132(23):2212-9. doi: 10.1161/CIRCULATIONAHA.115.017158. Epub 2015 Oct 5. PMID 26644246
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Schwingshackl L, Schwedhelm C, Galbete C, Hoffmann G. Adherence to Mediterranean Diet and Risk of Cancer: An Updated Systematic Review and Meta-Analysis. Nutrients. 2017 Sep 26;9(10):1063. doi: 10.3390/nu9101063. PMID 28954418
- [Background] Sotos-Prieto M, Bhupathiraju SN, Mattei J, Fung TT, Li Y, Pan A, Willett WC, Rimm EB, Hu FB. Association of Changes in Diet Quality with Total and Cause-Specific Mortality. N Engl J Med. 2017 Jul 13;377(2):143-153. doi: 10.1056/NEJMoa1613502. PMID 28700845
- [Background] Soltani S, Jayedi A, Shab-Bidar S, Becerra-Tomas N, Salas-Salvado J. Adherence to the Mediterranean Diet in Relation to All-Cause Mortality: A Systematic Review and Dose-Response Meta-Analysis of Prospective Cohort Studies. Adv Nutr. 2019 Nov 1;10(6):1029-1039. doi: 10.1093/advances/nmz041. PMID 31111871
- [Background] Delgado-Lista J, Alcala-Diaz JF, Torres-Pena JD, Quintana-Navarro GM, Fuentes F, Garcia-Rios A, Ortiz-Morales AM, Gonzalez-Requero AI, Perez-Caballero AI, Yubero-Serrano EM, Rangel-Zuniga OA, Camargo A, Rodriguez-Cantalejo F, Lopez-Segura F, Badimon L, Ordovas JM, Perez-Jimenez F, Perez-Martinez P, Lopez-Miranda J; CORDIOPREV Investigators. Long-term secondary prevention of cardiovascular disease with a Mediterranean diet and a low-fat diet (CORDIOPREV): a randomised controlled trial. Lancet. 2022 May 14;399(10338):1876-1885. doi: 10.1016/S0140-6736(22)00122-2. Epub 2022 May 4. PMID 35525255
- [Background] Kraus WE, Powell KE, Haskell WL, Janz KF, Campbell WW, Jakicic JM, Troiano RP, Sprow K, Torres A, Piercy KL; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Physical Activity, All-Cause and Cardiovascular Mortality, and Cardiovascular Disease. Med Sci Sports Exerc. 2019 Jun;51(6):1270-1281. doi: 10.1249/MSS.0000000000001939. PMID 31095084
- [Background] Aude YW, Agatston AS, Lopez-Jimenez F, Lieberman EH, Marie Almon, Hansen M, Rojas G, Lamas GA, Hennekens CH. The national cholesterol education program diet vs a diet lower in carbohydrates and higher in protein and monounsaturated fat: a randomized trial. Arch Intern Med. 2004 Oct 25;164(19):2141-6. doi: 10.1001/archinte.164.19.2141. PMID 15505128
- [Background] Diaz-Gutierrez J, Ruiz-Canela M, Gea A, Fernandez-Montero A, Martinez-Gonzalez MA. Association Between a Healthy Lifestyle Score and the Risk of Cardiovascular Disease in the SUN Cohort. Rev Esp Cardiol (Engl Ed). 2018 Dec;71(12):1001-1009. doi: 10.1016/j.rec.2017.10.038. Epub 2017 Dec 26. English, Spanish. PMID 29287797
- [Background] Li Y, Schoufour J, Wang DD, Dhana K, Pan A, Liu X, Song M, Liu G, Shin HJ, Sun Q, Al-Shaar L, Wang M, Rimm EB, Hertzmark E, Stampfer MJ, Willett WC, Franco OH, Hu FB. Healthy lifestyle and life expectancy free of cancer, cardiovascular disease, and type 2 diabetes: prospective cohort study. BMJ. 2020 Jan 8;368:l6669. doi: 10.1136/bmj.l6669. PMID 31915124
- [Background] Sotos-Prieto M, Moreno-Franco B, Ordovas JM, Leon M, Casasnovas JA, Penalvo JL. Design and development of an instrument to measure overall lifestyle habits for epidemiological research: the Mediterranean Lifestyle (MEDLIFE) index. Public Health Nutr. 2015 Apr;18(6):959-67. doi: 10.1017/S1368980014001360. Epub 2014 Jul 15. PMID 25025396
- [Background] Sotos-Prieto M, Santos-Beneit G, Bodega P, Pocock S, Mattei J, Penalvo JL. VALIDATION OF A QUESTIONNAIRE TO MEASURE OVERALL MEDITERRANEAN LIFESTYLE HABITS FOR RESEARCH APPLICATION: THE MEDITERRANEAN LIFESTYLE INDEX (MEDLIFE). Nutr Hosp. 2015 Sep 1;32(3):1153-63. doi: 10.3305/nh.2015.32.3.9387. PMID 26319833
- [Background] Pavicic Zezelj S, Kendel Jovanovic G, Kresic G. The association between the Mediterranean diet and high physical activity among the working population in Croatia. Med Pr. 2019 Apr 19;70(2):169-176. doi: 10.13075/mp.5893.00773. Epub 2019 Feb 21. PMID 30793709
- [Background] Hershey MS, Fernandez-Montero A, Sotos-Prieto M, Kales S, Gea A, Ruiz-Estigarribia L, Sanchez-Villegas A, Diaz-Gutierrez J, Martinez-Gonzalez MA, Ruiz-Canela M. The Association Between the Mediterranean Lifestyle Index and All-Cause Mortality in the Seguimiento Universidad de Navarra Cohort. Am J Prev Med. 2020 Dec;59(6):e239-e248. doi: 10.1016/j.amepre.2020.06.014. Epub 2020 Nov 18. PMID 33220762
- [Background] Mata-Fernandez A, Hershey MS, Pastrana-Delgado JC, Sotos-Prieto M, Ruiz-Canela M, Kales SN, Martinez-Gonzalez MA, Fernandez-Montero A. A Mediterranean lifestyle reduces the risk of cardiovascular disease in the "Seguimiento Universidad de Navarra" (SUN) cohort. Nutr Metab Cardiovasc Dis. 2021 Jun 7;31(6):1728-1737. doi: 10.1016/j.numecd.2021.02.022. Epub 2021 Feb 27. PMID 33895077
- [Background] Sotos-Prieto M, Ortola R, Ruiz-Canela M, Garcia-Esquinas E, Martinez-Gomez D, Lopez-Garcia E, Martinez-Gonzalez MA, Rodriguez-Artalejo F. Association between the Mediterranean lifestyle, metabolic syndrome and mortality: a whole-country cohort in Spain. Cardiovasc Diabetol. 2021 Jan 5;20(1):5. doi: 10.1186/s12933-020-01195-1. PMID 33402187
- [Background] Hershey MS, Sanchez-Villegas A, Sotos-Prieto M, Fernandez-Montero A, Pano O, Lahortiga-Ramos F, Martinez-Gonzalez MA, Ruiz-Canela M. The Mediterranean Lifestyle and the Risk of Depression in Middle-Aged Adults. J Nutr. 2022 Jan 11;152(1):227-234. doi: 10.1093/jn/nxab333. PMID 34549288
- [Background] Hershey MS, Sotos-Prieto M, Ruiz-Canela M, Christophi CA, Moffatt S, Martinez-Gonzalez MA, Kales SN. The Mediterranean lifestyle (MEDLIFE) index and metabolic syndrome in a non-Mediterranean working population. Clin Nutr. 2021 May;40(5):2494-2503. doi: 10.1016/j.clnu.2021.03.026. Epub 2021 Mar 31. PMID 33932793
- [Background] Maroto-Rodriguez J, Delgado-Velandia M, Ortola R, Garcia-Esquinas E, Martinez-Gomez D, Struijk EA, Lopez-Garcia E, Rodriguez-Artalejo F, Sotos-Prieto M. A Mediterranean Lifestyle and Frailty Incidence in Older Adults: The Seniors-ENRICA-1 Cohort. J Gerontol A Biol Sci Med Sci. 2022 Sep 1;77(9):1845-1852. doi: 10.1093/gerona/glab292. PMID 34614144
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937